CLINICAL TRIAL: NCT04371965
Title: Povidone Iodine Mouthwash, Gargle, and Nasal Spray to Reduce Naso- Pharyngeal Viral Load in Patients With SARS-CoV-2
Brief Title: Povidone Iodine Mouthwash, Gargle, and Nasal Spray to Reduce Naso- Pharyngeal Viral Load in Patients With COVID-19
Acronym: KILLER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KILLER
Record Dates: First submitted 2020-04-29; First posted 2020-05-01 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-07

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; Povidone Iodine decolonization
MeSH Terms: conditions — COVID-19 | interventions — Povidone-Iodine

STUDY DESIGN:
Intervention Model Description: Randomized controlled open label trial, parallel design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decolonization (Experimental): 1% Povidone iodine mouthwash (95 mL), gargle, and nasal spray (2,5 mL by nostril), and 10% nasal gel (one drop). All four time a day for five days.
  Interventions: Drug: Povidone-Iodine
- Control (No Intervention): Absence of local decolonization

INTERVENTIONS:
Drug: Povidone-Iodine — Patients in the experimental group will be asked to gargle with a 1% povidone-iodine solution, spray their nose with the same antiseptic solution, and finally applied 10% povidone-iodine cream in each nostril, all four times a day for five days.
  Arms: Decolonization

SUMMARY:
The SARS-CoV-2 coronavirus pandemic is responsible for more than 180,000 deaths worldwide and 20,000 deaths in France. To date, no treatment or vaccine has been successful. Povidone-iodine is an antiseptic suitable for use on the skin and mucosa with potent virucidal activity, particularly against coronaviruses. It is marketed for oro-nasopharyngeal decolonization.

24 patients with positive nasopharyngeal SARS-CoV-2 carriage will be randomized (1:1) in an experimental group (benefiting from povidone iodine decolonization) or a control group. Patients in the experimental group will be asked to gargle with a 1% povidone-iodine solution, spray their nose with the same antiseptic solution, and finally applied 10% povidone-iodine cream in each nostril, all four times a day for five days. Patients will be followed for 7 days to evaluate the efficacy and safety of povidone iodine decolonization.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age over 18 yrs) of both sexes
* With positive SARS-CoV-2 carriage by RT-PCR
* Having given their written consent after having been informed

Exclusion Criteria

* Patient with low viral load (threshold cycle [Ct] > 25 per RT-PCR),
* Patient unable to perform oro-nasopharyngeal decolonization
* Known hypersensitivity to one of the constituents, particularly to povidone-iodine,
* History of dysthyroidism,
* Known coagulopathy,
* Participation in another clinical trial aimed at reducing viral load in patients with SARS-CoV-2,
* Pregnant or breastfeeding women, or women of childbearing age without effective contraception
* Patients not covered by a social security scheme
* Patients with enhanced protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-10-23 (Actual); Study Completion 2020-10-23 (Actual)

PRIMARY OUTCOMES:
Change from baseline naso-pharyngeal viral load quantified by RT-PCR at Day7 | Day 7

SECONDARY OUTCOMES:
Delay between inclusion and negativation of SARS-CoV-2 nasopharyngeal carriage | Day0, Day1, Day3, Day5 and Day7
Delay between inclusion and negativation of SARS-CoV-2 nasopharyngeal cell cultures | Day0, Day1, Day3, Day5 and Day7
Thyroid tests at Day0 and Day7 | Day0 and Day7
Patient satisfaction at Day7 using a numerical comfort scale, graduated from 0 (any discomfort) to 10 (maximum possible discomfort) | Day7
Daily presence of clinical signs in favour of COVID-19, including respiratory distress using NYHA scale, chest pain, anosmia, agueusia, tiredness, cough, stiffness, nasal congestion, dysphagia and diarrhea | Day0, Day1, Day3, Day5 and Day7
Need for ward or intensive care hospitalization | Day0, Day1, Day3, Day5 and Day7

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Poitiers, Poitiers, France

REFERENCES:
- [Derived] Guenezan J, Garcia M, Strasters D, Jousselin C, Leveque N, Frasca D, Mimoz O. Povidone Iodine Mouthwash, Gargle, and Nasal Spray to Reduce Nasopharyngeal Viral Load in Patients With COVID-19: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2021 Apr 1;147(4):400-401. doi: 10.1001/jamaoto.2020.5490. PMID 33538761